CLINICAL TRIAL: NCT03846973
Title: Evaluation of the Safety and Efficacy of the Second Dose of Tranexamic Acid Administration of Trauma Patients: A Randomized, Double-blind Controlled Clinical Trial
Brief Title: Evaluation of the Safety and Efficacy of the Second Dose of Tranexamic Acid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Ayman El-Menyar, Director, Trauma & Vascular Research, Hamad Medical Corporation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16417/16
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Tranexamic Acid
Keywords: Trauma, Mortality, Tranexamic , Prehospital
MeSH Terms: conditions — Wounds and Injuries | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tranexamic acid (Experimental): group-I will include 110 patients with initial pre-hospital TXA administered slowly over 10 minutes followed by an intravenous infusion of 1 g TXA to be given and completed over 8 h in the hospital
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): group-II will include 110 patients with initial pre-hospital TXA administered slowly over 10 minutes but will receive placebo (normal saline) infusion to be given and completed over 8 h in the hospital
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — intravenous infusion of 1 g infusion to be given and completed over 8 h in the hospital
  Other Names: TXA
  Arms: Tranexamic acid
Other: Placebo — placebo (normal saline) infusion to be given and completed over 8 h in the hospital
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
TXA is currently administered pre-hospital in Canada, Germany, United Kingdom and Israel . These studies demonstrated that TXA use did not result in any detectable complications or adverse events. It is considered an ideal pre-hospital treatment because: (a) patients with severe hemorrhage die early more often than patients without hemorrhage; (b) it seems that the earlier treatment is administered, the better; (c) it is stable and easily stored; and (d) it is easily administered by paramedics. Herein, the study aimed to evaluate the effect of administration of second dose of Tranexamic acid infusion in the hospital setting in comparison to not receiving the second dose on the outcomes of trauma patients with an evidence of significant hemorrhage.

Recently, HGH ambulance service has included pre-hospital administration of TXA in trauma patients with significant hemorrhage. So, all eligible trauma patients will receive pre-hospital TXA (first dose) slowly over 10 minutes by the critical care paramedics as standard of care.

Inclusion Criteria: All adult trauma male and female patients (≥18 or <90 years) with evidence of significant hemorrhage (systolic blood pressure <90 mmHg or heart rate >110 beats per minutes, or both) or had Capillary Refill Time 3-4 seconds and received first dose of prehospital TXA will be included in the study.

Exclusion criteria:

1. Age > 90 or < 18 years of age
2. Inability to obtain intravenous access (intraosseous access not sufficient)
3. Documented cervical cord injury with motor deficit
4. Known prisoner
5. Known pregnancy
6. Traumatic arrest with > 5 minutes CPR without return of vital signs
7. Penetrating cranial injury
8. Traumatic brain injury with brain matter exposed
9. Isolated drowning or hanging victims
10. Wearing an opt out bracelet. Patient data will include demographics, time since injury, type of injury (blunt or penetrating), Glasgow Coma Score(GCS), Injury severity score (ISS), systolic blood pressure, respiratory rate, central capillary refill time, estimated number of hours since injury, laboratory findings, blood transfusion, units of transfused blood, management, complications and outcome.

The primary outcome will be death in hospital within 4 weeks of injury. Secondary outcomes will be morbidity (thromboembolic events, sepsis, Acute respiratory distress syndrome and organ failure), and number of blood transfusions (Massive transfusion protocol) and hospital length of stay.

DETAILED DESCRIPTION:
Study design It is a single-center, prospective, double-blind, randomized, placebo-controlled trial.

Study population All severely injured male and female patients with evidence of significant hemorrhage (systolic blood pressure <90 mmHg or heart rate >110 beats per minutes, or both) or had Capillary Refill Time 3-4 seconds will be administered TXA slowly over 10 minutes at the prehospital settings by critical care paramedics as standard of care are eligible for participation in this trial.

Sample size estimation:

The present clinical trial is based on CRASH-2 study [2] in which the sample size was more than 20,000 using the followings primary outcomes estimates such as all-cause-mortality 14.5% (TXA) vs. 16% (Placebo) and bleeding: 4.9% (TXA) vs. 5.7% (Placebo). According to CRASH-2 study approximately 30% of all patients randomized presented with significant hypotension (blood pressure < 90 mm Hg) considered to have significant hemorrhage.

This is a unique study to assess the effect of second dose of tranexamic acid in the hospital setting and there are no precise estimates available on the primary outcome particularly in our population. According to CRASH-2 trial, approximately 30% of all randomized patients presented with significant hypotension (BP <90mmHg) indicated hemorrhagic shock. Therefore, taking the prevalence of hemorrhage to be 30% with 5% confidence limit and 80% power; a total of 335 trauma patients need to be included in the study.

There will be three arms in this trial; Group-1 will include 110 patients with initial pre-hospital TXA administered slowly over 10 minutes followed by in-hospital intravenous infusion of 1 g TXA administer over 8 h; Group-2 will include 110 patients with initial pre-hospital TXA administered slowly over 10 minutes but will receive placebo over 8 h in the hospital and Group-3 will include 110 age and injury severity score (ISS) matched historical controls without TXA administration identified from hospital database (January 1, 2016 till December 31, 2016).

Each study package will be labelled with the study protocol number, unique randomization code, and name of the principal investigator. All study treatment pack will contain two ampules of either tranexamic acid 500 mg or placebo, one 100 ml bag of 0.9% saline, a syringe and needle, stickers with the trial details and randomization number (for attaching to infusion bags, data forms, and patient medical records), and instructions. Each box contained information leaflets for patients and their representatives, consent forms, and data collection forms. The stickers, instructions, leaflets, and forms will be available in English and Arabic. A small number of details will be completed on the wristband and label (Patient's initials, Date and time of randomization). The label will be placed in the patient's hospital medical record. The wristband and label in the patient's medical record will alert hospital staff to the patient's enrollment in the study. The principal investigator or their designee is responsible for ensuring the drug or placebo is administered according to the study protocol and they will be unaware of whether the patient was assigned to the TXA or placebo group.

The research team including research coordinator will be notified by the treating physician about the recruitment. Detailed interventions are mentioned in study procedures below.

10 ml blood specimen will be drawn for coagulation profile (INR, PT, PTT, Fibrinogen, and D-Dimer); 5 ml before and 5 ml after starting TXA. The data will be collected prospectively with the help of a predesigned data collection form. Patient data included sex, age, nationality, time since injury, type of injury (blunt or penetrating), Glasgow Coma Score(GCS), Injury severity score (ISS), systolic blood pressure, respiratory rate, central capillary refill time, estimated number of hours since injury, laboratory findings, blood transfusion, units of transfused blood, management, complications and outcome.

The primary outcome will be death in hospital within 4 weeks of injury. Secondary outcomes will be morbidity (thromboembolic events, sepsis, Acute respiratory distress syndrome and organ failure), and number of blood transfusions (Massive transfusion protocol) and hospital length of stay.

Study Population Pre-hospital administration of TXA in trauma patients with evidence of significant hemorrhage is being included in the HGH ambulance service. So, all eligible trauma patients with risk of bleeding will receive pre-hospital TXA slowly over 10 minutes by the critical care paramedics as standard of care. In the hospital, subjects will be assessed by study trained treating physician and if they fulfill the inclusion criteria and have no exclusion criteria they will be randomized to give second 8-hour infusion of TXA or placebo by opening the next opaque envelope in the randomization series. The envelopes will contain a wristband to be placed on the patient & a label which designates the study number and treatment allocation. A small number of details will be completed on the wristband and label (patient's initials, date and time of randomization). The label will be placed in the patient's hospital medical record. The wristband and label in the patient's medical record will alert hospital staff to the patient's enrollment in the study.

The research team including research coordinator will be notified by the treating physician about the recruitment.

The information regarding patient's enrollment will be kept confidential and all study related steps (explanation of study procedures and consenting) with the next of kin will be done in isolated room in the emergency area to maintain complete privacy. No one outside the research team and next of kin will be aware about the patient's participation in the study.

Recruited subjects will receive a specific study number. The research coordinator will compile a study enrollment log which will link the study number to the patient's details. Subsequent data will be identified by the study number. The enrollment log and study data will be kept separately. All data collected for the assessment will be identified by the study code. Study data will be entered into a password protected computer with study documents will be kept in a locked office with principal investigator at HMC.

Study drug Each 5 mL ampule contains 500 gm (×2) tranexamic acid and 10 mL water for injection as the inactive ingredient. Tranexamic acid solution for injection is a sterile, clear, colorless solution. The pH is 6.5 to 8.0. The placebo is identical in appearance and packaging but contains sodium chloride 0.9% w/v in a 10 mL ampule.

It is a randomized double blind placebo controlled single center trial. Eligible subjects will be screened and enrolled in the hospital by the treating physician. If they fulfill the inclusion criteria and have no exclusion criteria they will be randomized into either of the group (Group-1 or group-2) by opening the next opaque envelope in the randomization series kept in the trauma room. The envelopes will contain a wristband to be placed on the patient & a label which designates the study number and treatment. A small number of details will be completed on the wristband and label (Patient's initials, Date and time of randomization). The label will be placed in the patient's hospital electronic medical record. The wristband and label in the patient's medical record will alert hospital staff to the patient's enrollment in the study.

Blinding Blinding will be done through pharmacy department where both tranexamic acid and normal saline will be placed in similar bags in IV admixture room, both are colorless. Total of 220 bags will be numbered, the codes will be kept confidential and not broken unless emergency case.

The emergency physicians will be unable to determine whether a trial pack contains the active study drug or placebo as they are both identical in appearance. The unique study ID number printed on the trial pack and the contents within the pack is the only way to determine whether a pack contains active drug or placebo. The coded list of study ID numbers is only accessible to the independent study coordinator and will not be accessible to researchers involved in the trial until after the trial is completed (individual cases may be unblinded in exceptional circumstances as per emergency unblinding mentioned below). Both participants and study staff (investigators and trial staff) will be masked to treatment allocation.

Emergency unblinding

The treating physician at emergency department will ask for unblinding for the sake of patient care, if unblinding is needed based on the clinical progress of the patient following steps will be followed:

Procedure for emergency unblinding:

1. In case of emergency, the treating physician will contact the trial coordinator to break the code.
2. The trial coordinator will provide with the information as requested.
3. The study code should only be broken when the treating physician believes that clinical management depends importantly upon knowledge of whether the patient received antifibrinolytic or placebo. In those few cases only, unblinding will be allowed to know whether the patient received antifibrinolytic or placebo.
4. On receipt of the treatment allocation details, treating physician deals with the participant's medical emergency as appropriate.
5. If the treating physician is not the PI, the treating physician must inform the PI of the code break and the reasons for the actions taken as soon as possible.
6. The PI documents the breaking of the code and the reasons for doing so on the data collection sheet.
7. The PI documents the breaking of the codes in a separate file. Discontinuation of treatment Study medication will be ceased permanently for any occurrence of serious adverse event such as seizure, cardiac arrest or anaphylaxis. Ultimately the treating clinician will have the right to decide whether to discontinue treatment, ideally this should be discussed with the principal investigator where feasible. All patients with discontinued treatment of the study drug will be followed for outcomes.

Significance This trial aims to determine the overall benefits and harms of giving second infusion of TXA for severely injured patients in the emergency room. Importantly, it aims to determine whether TXA infusion as compared to single dose will affect the outcomes of the trauma patients with significant bleeding. It is timely that it will objectively resolve current uncertainty about whether the benefits of TXA infusion versus single dose will outweigh any potential harm for severely injured patients in prehospital setting in our region. The potential benefit of TXA to significantly improve mortality rates and secondary outcomes for patients could result in significant savings in lifetime costs and improved quality of life following severe injury. If this trial proves a beneficial effect of early TXA infusion of second dose of TXA in hospital setting in terms of outcomes, than it will be used for all trauma patients with significant bleeding. On the other hand, if single dose shows similar benefit in terms of outcomes than it can mitigate the side effects that could be raised with the second dose of TXA infusion and would recommend using only single dose of TXA in the prehospital settings. Finally, this trial will demonstrate the ability of our trauma services to appropriately select patients and administer a time-critical drug treatment to minimize harmful consequences of hemorrhage in major trauma.

ELIGIBILITY:
Inclusion Criteria:

All adult trauma male and female patients (≥18 or <90 years) with evidence of significant hemorrhage (systolic blood pressure <90 mmHg or heart rate >110 beats per minutes, or both) or had Capillary Refill Time 3-4 seconds [2] and received first dose of prehospital TXA will be included in the study.

Exclusion Criteria:

1. Age > 90 or < 18 years of age
2. Inability to obtain intravenous access (intraosseous access not sufficient)
3. Documented cervical cord injury with motor deficit
4. Known prisoner
5. Known pregnancy
6. Traumatic arrest with > 5 minutes CPR without return of vital signs
7. Penetrating cranial injury
8. Traumatic brain injury with brain matter exposed
9. Isolated drowning or hanging victims
10. Wearing an opt out bracelet.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2018-12-02 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
mortality | 4 weeks post injury
  Number of participants who died from each study arm

SECONDARY OUTCOMES:
morbidity | 4 weeks post injury
  Number of participants of each study arm who developed thromboembolic events, sepsis, Acute respiratory distress syndrome and organ failure)
number of blood transfusions | 4 weeks post injury
  number of participants of each study arm who received blood transfusions (MTP: massive transfusion protocol)
Hospital length of stay | 4 weeks post injury
  Number of hospital length of stay for each study group

CONTACTS AND LOCATIONS:
Locations (1):
- Hamad General Hospital, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No
Only the lead PI will have the access to the data which will be coded with subject identifier to ensure data safety and confidentiality.

REFERENCES:
- [Background] Asim M, El-Menyar A, Al-Thani H, Abdelrahman H, Zarour A, Latifi R. Blunt traumatic injury in the Arab Middle Eastern populations. J Emerg Trauma Shock. 2014 Apr;7(2):88-96. doi: 10.4103/0974-2700.130878. PMID 24812453
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] World Health Organization. Violence, Injuries, and Disability: Biennial 2008-2009 Report. Geneva, Switzerland: WHO; 2010.
- [Background] Sauaia A, Moore FA, Moore EE, Moser KS, Brennan R, Read RA, Pons PT. Epidemiology of trauma deaths: a reassessment. J Trauma. 1995 Feb;38(2):185-93. doi: 10.1097/00005373-199502000-00006. PMID 7869433
- [Background] Heckbert SR, Vedder NB, Hoffman W, Winn RK, Hudson LD, Jurkovich GJ, Copass MK, Harlan JM, Rice CL, Maier RV. Outcome after hemorrhagic shock in trauma patients. J Trauma. 1998 Sep;45(3):545-9. doi: 10.1097/00005373-199809000-00022. PMID 9751548
- [Background] Brohi K, Cohen MJ, Ganter MT, Schultz MJ, Levi M, Mackersie RC, Pittet JF. Acute coagulopathy of trauma: hypoperfusion induces systemic anticoagulation and hyperfibrinolysis. J Trauma. 2008 May;64(5):1211-7; discussion 1217. doi: 10.1097/TA.0b013e318169cd3c. PMID 18469643
- [Background] Hess JR, Brohi K, Dutton RP, Hauser CJ, Holcomb JB, Kluger Y, Mackway-Jones K, Parr MJ, Rizoli SB, Yukioka T, Hoyt DB, Bouillon B. The coagulopathy of trauma: a review of mechanisms. J Trauma. 2008 Oct;65(4):748-54. doi: 10.1097/TA.0b013e3181877a9c. PMID 18849786
- [Background] Brohi K, Singh J, Heron M, Coats T. Acute traumatic coagulopathy. J Trauma. 2003 Jun;54(6):1127-30. doi: 10.1097/01.TA.0000069184.82147.06. PMID 12813333
- [Background] Hoylaerts M, Lijnen HR, Collen D. Studies on the mechanism of the antifibrinolytic action of tranexamic acid. Biochim Biophys Acta. 1981 Feb 18;673(1):75-85. No abstract available. PMID 7193484
- [Background] Henry DA, Moxey AJ, Carless PA, O'Connell D, McClelland B, Henderson KM, Sly K, Laupacis A, Fergusson D. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2001;(1):CD001886. doi: 10.1002/14651858.CD001886. PMID 11279735
- [Background] Horrow JC, Hlavacek J, Strong MD, Collier W, Brodsky I, Goldman SM, Goel IP. Prophylactic tranexamic acid decreases bleeding after cardiac operations. J Thorac Cardiovasc Surg. 1990 Jan;99(1):70-4. PMID 2403616
- [Background] Horrow JC, Van Riper DF, Strong MD, Brodsky I, Parmet JL. Hemostatic effects of tranexamic acid and desmopressin during cardiac surgery. Circulation. 1991 Nov;84(5):2063-70. doi: 10.1161/01.cir.84.5.2063. PMID 1934382
- [Background] Boylan JF, Klinck JR, Sandler AN, Arellano R, Greig PD, Nierenberg H, Roger SL, Glynn MF. Tranexamic acid reduces blood loss, transfusion requirements, and coagulation factor use in primary orthotopic liver transplantation. Anesthesiology. 1996 Nov;85(5):1043-8; discussion 30A-31A. doi: 10.1097/00000542-199611000-00012. PMID 8916821
- [Background] Zufferey PJ, Miquet M, Quenet S, Martin P, Adam P, Albaladejo P, Mismetti P, Molliex S; tranexamic acid in hip-fracture surgery (THIF) study. Tranexamic acid in hip fracture surgery: a randomized controlled trial. Br J Anaesth. 2010 Jan;104(1):23-30. doi: 10.1093/bja/aep314. PMID 19926634
- [Background] Lawson JH, Murphy MP. Challenges for providing effective hemostasis in surgery and trauma. Semin Hematol. 2004 Jan;41(1 Suppl 1):55-64. doi: 10.1053/j.seminhematol.2003.11.012. PMID 14872423
- [Background] Henry DA, Carless PA, Moxey AJ, O'Connell D, Stokes BJ, Fergusson DA, Ker K. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2011 Mar 16;2011(3):CD001886. doi: 10.1002/14651858.CD001886.pub4. PMID 21412876
- [Background] Levy JH. Antifibrinolytic therapy: new data and new concepts. Lancet. 2010 Jul 3;376(9734):3-4. doi: 10.1016/S0140-6736(10)60939-7. Epub 2010 Jun 14. No abstract available. PMID 20554318
- [Background] CRASH-2 collaborators; Roberts I, Shakur H, Afolabi A, Brohi K, Coats T, Dewan Y, Gando S, Guyatt G, Hunt BJ, Morales C, Perel P, Prieto-Merino D, Woolley T. The importance of early treatment with tranexamic acid in bleeding trauma patients: an exploratory analysis of the CRASH-2 randomised controlled trial. Lancet. 2011 Mar 26;377(9771):1096-101, 1101.e1-2. doi: 10.1016/S0140-6736(11)60278-X. PMID 21439633
- [Background] Morrison JJ, Dubose JJ, Rasmussen TE, Midwinter MJ. Military Application of Tranexamic Acid in Trauma Emergency Resuscitation (MATTERs) Study. Arch Surg. 2012 Feb;147(2):113-9. doi: 10.1001/archsurg.2011.287. Epub 2011 Oct 17. PMID 22006852
- [Background] Inaba K. Antifibrinolytics in trauma patients: does it MATTER? Arch Surg. 2012 Feb;147(2):119. doi: 10.1001/archsurg.2011.286. Epub 2011 Oct 17. No abstract available. PMID 22351905
- [Background] Vu EN, Schlamp RS, Wand RT, Kleine-Deters GA, Vu MP, Tallon JM. Prehospital use of tranexamic acid for hemorrhagic shock in primary and secondary air medical evacuation. Air Med J. 2013 Sep-Oct;32(5):289-92. doi: 10.1016/j.amj.2013.05.001. PMID 24001917
- [Background] Lipsky AM, Abramovich A, Nadler R, Feinstein U, Shaked G, Kreiss Y, Glassberg E. Tranexamic acid in the prehospital setting: Israel Defense Forces' initial experience. Injury. 2014 Jan;45(1):66-70. doi: 10.1016/j.injury.2013.08.025. Epub 2013 Sep 7. PMID 24074828
- [Background] Wafaisade A, Lefering R, Bouillon B, Bohmer AB, Gassler M, Ruppert M; TraumaRegister DGU. Prehospital administration of tranexamic acid in trauma patients. Crit Care. 2016 May 12;20(1):143. doi: 10.1186/s13054-016-1322-5. PMID 27176727
- [Background] Paudyal P, Smith J, Robinson M, South A, Higginson I, Reuben A, Shaffee J, Black S, Logan S. Tranexamic acid in major trauma: implementation and evaluation across South West England. Eur J Emerg Med. 2017 Feb;24(1):44-48. doi: 10.1097/MEJ.0000000000000323. PMID 26313316
- [Background] Pre-hospital Anti-fibrinolytics for Traumatic Coagulopathy and Haemorrhage (The PATCH Study) (PATCH). Ongoing Clinical Trials. Retrieved from https://clinicaltrials.gov/ct2/show/NCT02187120 accessed on May 20, 2016
- [Background] Apodaca A, Olson CM Jr, Bailey J, Butler F, Eastridge BJ, Kuncir E. Performance improvement evaluation of forward aeromedical evacuation platforms in Operation Enduring Freedom. J Trauma Acute Care Surg. 2013 Aug;75(2 Suppl 2):S157-63. doi: 10.1097/TA.0b013e318299da3e. PMID 23883901
- [Background] Glassberg E, Nadler R, Gendler S, Abramovich A, Spinella PC, Gerhardt RT, Holcomb JB, Kreiss Y. Freeze-dried plasma at the point of injury: from concept to doctrine. Shock. 2013 Dec;40(6):444-50. doi: 10.1097/SHK.0000000000000047. PMID 24089000
- [Background] Ausset S, Glassberg E, Nadler R, Sunde G, Cap AP, Hoffmann C, Plang S, Sailliol A. Tranexamic acid as part of remote damage-control resuscitation in the prehospital setting: A critical appraisal of the medical literature and available alternatives. J Trauma Acute Care Surg. 2015 Jun;78(6 Suppl 1):S70-5. doi: 10.1097/TA.0000000000000640. PMID 26002268
- [Background] Neeki MM, Dong F, Toy J, Vaezazizi R, Powell J, Jabourian N, Jabourian A, Wong D, Vara R, Seiler K, Pennington TW, Powell J, Yoshida-McMath C, Kissel S, Schulz-Costello K, Mistry J, Surrusco MS, O'Bosky KR, Van Stralen D, Ludi D, Sporer K, Benson P, Kwong E, Pitts R, Culhane JT, Borger R. Efficacy and Safety of Tranexamic Acid in Prehospital Traumatic Hemorrhagic Shock: Outcomes of the Cal-PAT Study. West J Emerg Med. 2017 Jun;18(4):673-683. doi: 10.5811/westjem.2017.2.32044. Epub 2017 Apr 19. PMID 28611888
- [Background] Huebner BR, Dorlac WC, Cribari C. Tranexamic Acid Use in Prehospital Uncontrolled Hemorrhage. Wilderness Environ Med. 2017 Jun;28(2S):S50-S60. doi: 10.1016/j.wem.2016.12.006. PMID 28601210
- [Background] Electronics Medicines Compendium (2011) Cyklopron Standard Product Characteristics. http://www.medicines.org.uk/EMC/medicine/1489/SPC/Cyklokapron+Injection/ [Accessed 23rd May 2016].
- [Background] Guerriero C, Cairns J, Perel P, Shakur H, Roberts I; CRASH 2 trial collaborators. Cost-effectiveness analysis of administering tranexamic acid to bleeding trauma patients using evidence from the CRASH-2 trial. PLoS One. 2011 May 3;6(5):e18987. doi: 10.1371/journal.pone.0018987. PMID 21559279
- [Background] World Health Organisation (2011) Model Lists of Essential Medicines. 17th Ed. http://www.who.int/medicines/publications/essentialmedicines/en/ Accessed 23rd May 2016].
- [Derived] El-Menyar A, Ahmed K, Hakim S, Kanbar A, Mathradikkal S, Siddiqui T, Jogol H, Younis B, Taha I, Mahmood I, Ajaj A, Atique S, Alaieb A, Bahey AA, Asim M, Alinier G, Castle NR, Mekkodathil A, Rizoli S, Al-Thani H. Efficacy and safety of the second in-hospital dose of tranexamic acid after receiving the prehospital dose: double-blind randomized controlled clinical trial in a level 1 trauma center. Eur J Trauma Emerg Surg. 2022 Aug;48(4):3089-3099. doi: 10.1007/s00068-021-01848-0. Epub 2021 Dec 15. PMID 34910219